CLINICAL TRIAL: NCT03399279
Title: Comparative Study Of Perforated Versus Non Perforated Collagen Membrane Combined With Nanohydroxyapatite In The Management Of Intrabony Defects
Brief Title: Perforated Collagen Membrane With Nanohydroxyapatite for Intrabony Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hesham Mohammed Abdallah, Dr., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0925-0586
Record Dates: First submitted 2018-01-08; First posted 2018-01-16 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Intrabony Periodontal Defect
Keywords: nanohydroxyapatite; Perforated membrane; occlusive membrane; Aggressive periodontitis
MeSH Terms: conditions — Aggressive Periodontitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open flap debridement & perforated&Nano (Experimental): Perforated collagen membrane and nano-hydroxyapatite and open flap debridement
  Interventions: Procedure: Open flap debridment; Other: Perforated collagen membrane; Other: Nanohydroxyapetite
- Open flap debridment &Occlusive&Nano (Active Comparator): Occlusive membrane and nano-hydroxyapatite and open flap debridement
  Interventions: Procedure: Open flap debridment; Other: Occlusive membrane; Other: Nanohydroxyapetite

INTERVENTIONS:
Procedure: Open flap debridment — Full mucoperiosteal flap reflected+ Debridement of infrabony defect
Other: Perforated collagen membrane — Membrane perforations using dental needle
  Arms: Open flap debridement & perforated&Nano
Other: Occlusive membrane — Biotech collagen membrane
  Arms: Open flap debridment &Occlusive&Nano
Other: Nanohydroxyapetite — Nanbone Particles

SUMMARY:
The ultimate goal of periodontal therapy is the regeneration of periodontal tissues which have been destroyed due to periodontal disease. Different modalities have been proposed to obtain regeneration of periodontal tissues employing various bone grafts, bone substitute materials, guided tissue regeneration (GTR), combination of bone grafts or bone substitutes with GTR, and growth factors.

So, a new, fully synthetic, nanocrystalline, unsintered, phase-pure hydroxyapatite (nano-HA) has been suggested as a potential material for enhancing periodontal and bone regeneration since its chemical composition and crystalline structure correspond to the calcium phosphate component of natural bone and may have greater potential for resorption compared with sintered hydroxyapatite.

A study performed in 2012, on 14 patients with paired intrabony periodontal defects of ≥4 mm participated in split mouth design study. The defects in each subject were randomly selected to receive nano-HA paste in conjunction with papilla preservation flaps or papilla preservation flaps alone. Probing bone levels from a customized acrylic stent and probing pocket depths were measured at baseline and again 6 months following surgery. No differences in any of the investigated parameters were observed at baseline between the two groups. Healing was uneventful in all patients. Both treatments resulted in significant improvements between baseline and 6 months in all clinical and radio-graphic parameters. In conclusion, they found that the nano crystalline hydroxyapatite bone graft in combination with collagen membrane demonstrated clinical advantages beyond that achieved by open flap debridement alone.

The concept of porous guided tissue membrane has been tested recently as a modality that could stimulate bone formation of critical sized bone defects. Kim and co-workers claimed that asymmetrically porous GBR membranes with dual BMP-2 and ultrasound stimulation may be promising for the clinical treatment of delayed and insufficient bone healing. For guided tissue regeneration in periodontal therapy, membrane perforations could allow for gingival stem cells and periosteal cells to take part in supracrestal regeneration. The perforated section of the membranes would stabilize supracrestal fibrin clot through mechanical interlocking of fibrin strands with the membrane pores providing more membrane and clot stability. It has been suggested that regenerative failures may result when the tensile strength of the fibrin clot is exceeded, resulting in a tear and a long junctional epithelium type attachment.

DETAILED DESCRIPTION:
The study will be conducted on 12 individuals. The research esthetics committee of Faculty of Dentistry, Ain Shams University will review the proposal.

All patients will be informed about the nature of the study and will fine an informed consent.

I - Selection of the patients:

The patients will be selected from the outpatient clinic of Oral Medicine and Periodontology department, Faculty of Dentistry, Ain Shams University.

All the selected patients will be selected according to following criteria:

Inclusion criteria:

1. Patients free from any systemic diseases as evidenced by health using Burket's Oral Medicine health history questionnaire. (Glick, 2008)
2. Patients' age range from 25 to 50 years old.
3. Each patient should have at least two contralateral intrabony defects which fulfill the following criteria:

   (i) Probing depth ≥ 5 mm. (ii) Clinical attachment loss ≥ 5 mm. (iii) Radiographic evidence of vertical bone loss using periapical radiographs.
4. Patients are should be willing to participate in the study and should be able to return for the follow up visits.

Exclusion criteria:

1. Patients with history of periodontal surgery or medications including antibiotics and non-steroidal anti-inflammatory drugs for at least 3 months prior to the initiation of the study.
2. Pregnant females as well as breast feeding mothers.
3. Smokers.
4. Vulnerable groups as prisoners, mentally disabled, etc… All participants following initial clinical examination and periapical radiographs will be given detailed instructions in self-performed plaque control measures, including tooth brushing and dental flossing. All patients will receive full mouth scaling and root planing using ultra-sonic scalers and hand instruments under local anesthesia to minimize patient discomfort.

II- Study groups:

The selected sites will be randomly "double blinded study" divided into two groups in a split mouth design.

Group One:

The defects will be treated with open flap debridment followed by the placement of nanohydroxyapetite* combined with perforated collagen membrane**.

Group Two:

The defects will be treated with open flap debridment followed by the placement of nanohydroxyapetite combined with non perforated collagen membrane.

The mucoperiosteal flaps will be adapted and sutured and the patients will be given post-surgical instructions.

III- Periodontal evaluation:

Clinical Parameters:

The clinical parameters will be measured at one, three and six months postoperatively.

1) Plaque index (PI): Criteria of plaque index (PI) of (Silness and Loe, 1969) 0: No plaque in gingival area.

1. No plaque visible by the unaided eye, but plaque is made visible on the point of the probe after it has been moved across surface at entrance of gingival crevice.
2. Gingival area is covered with thin to moderately thick layer of plaque, deposit is visible to naked eye.
3. Heavy accumulation of plaque, the thickness of which fills out niche produced by gingival margin and tooth surface, inter dental area is stuffed with plaque.

2) Gingival index (GI): Criteria of the gingival index (GI) of (Loe, 1967) 0: Normal gingiva

1. Mild inflammation: slight change in color and slight edema; no bleeding on probing.
2. moderate inflammation: redness, edema and glazing; bleeding on probing.
3. Severe inflammation: marked redness and edema; ulceration; tendency to spontaneous bleeding.

3) Probing pocket depth (PPD) : Probing pocket depth (PPD) will be measured from the gingival margin to the base of periodontal pocket to the nearest mm (Caton, 1989).

Six readings will be recorded for each tooth: Mesiobuccal, mid-buccal, distobuccal, mesiolingual, mid-lingual and distolingual.

4) Clinical attachment level (CAL): Clinical attachment level will be measured from cementoenamel junction to the base of pocket to the nearest mm.

B- Radiographic parameters

Periapical radiographs and Cone beam computed tomography will be taken at base line and at six months after the placement of barrier membranes combined with nanohydroxyapatite and the following parameters will be measured:

The sites will be measured first on periapical radiographs and later on CBCT with the help of the ruler in the Image Tool software (University of Texas Health Science Centre, San Antonio, TX) based on the method proposed by Misch et al.

Three measurements will be performed for each site:

1. The height of the alveolar crest (AC): measured from the cementoenamel junction (CEJ) to the AC.
2. The depth of the defect, measured from the CEJ to the bottom of the defect.
3. The width of the defect, measured from the highest point of the AC to the dental root adjacent to the defect.

The axial slices will be used to verify the presence of combined bone defects and identify according to the classification of Goldman and Cohen.

ELIGIBILITY:
Inclusion Criteria:

* Patients free from any systemic diseases as evidenced by health using Burket's Oral Medicine health history questionnaire. (Glick, 2008)
* Patients' age range from 25 to 50 years old.
* Each patient should have at least two contralateral intrabony defects which fulfill the following criteria: ** Probing depth ≥ 5 mm.

  * Clinical attachment loss ≥ 5 mm.
  * Radiographic evidence of vertical bone loss using periapical radiographs.
* Patients are should be willing to participate in the study and should be able to return for the follow up visits.

Exclusion Criteria:

* Patients with history of periodontal surgery or medications including antibiotics and non-steroidal anti-inflammatory drugs for at least 3 months prior to the initiation of the study.
* Pregnant females as well as breast feeding mothers.
* Smokers.
* Vulnerable groups as prisoners, mentally disabled, etc…

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2014-12-17 (Actual); Primary Completion 2016-09-15 (Actual); Study Completion 2017-03-25 (Actual)

PRIMARY OUTCOMES:
CAL | Change from base line to 3 months and 6 months
  Clinical attachment level

SECONDARY OUTCOMES:
DOD | Change from base line to 6 months
  Depth of Defect (From cemento enamel junction to defect base)